CLINICAL TRIAL: NCT01463761
Title: Autonomic Nervous System, Fatigue and Intolerance to Physical Training, and Overtraining in High-Level Athletes. A Multicentre Study
Brief Title: Autonomic Nervous System, Fatigue and Intolerance to Physical Training, and Overtraining in High-Level Athletes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Minister of Youth Affairs and Sports, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0908073; 2009-A00674-53 (Other: AFSSAPS)
Record Dates: First submitted 2011-10-31; First posted 2011-11-02 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Athletes; Training; Fatigue
Keywords: High-level athlete; ANS activity; Overtraining
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- high-level athletes: High-level athlete, enrolled in a Ministry-recognized Pôle
  Interventions: Device: ANS activity

INTERVENTIONS:
Device: ANS activity — This ANS activity is measured by nocturnal heart rates records with Holter ECG.

SUMMARY:
Sports training aims to enhance an athlete's performance (overcompensation). To do that, the athlete must go through periods of fatigue and lower performance (overreaching). When the training plan is balanced, this fatigue is short and reversible.If the training load is too heavy or if recuperation periods are too short, it can lead to persistence fatigue that may only be reversible in the long term. This state of fatigue is part of the broader clinical picture of overtraining, which includes stark changes in performance as well as mood and sleep disorders. Many prediction and characterization methods based on biological markers have been evaluated, but they have not been put into practice in sports training due to obstacles such as reliability, interindividual variability and high costs. This study aims to evaluate a new approach based on the variability of an individual's heart rate (RR variability), which is a way of measuring autonomic nervous system (ASN) activity. It is non-invasive, low-cost, and has already proven useful in athlete health monitoring.

DETAILED DESCRIPTION:
The investigators propose to describe the variation of these ANS regulation factors over a full year, in a population of high-level athletes, in order to measure changes in regulation which may be predictive of potential fatigue and intolerance to physical training, if such a syndrome came to be observed among the study group.

ELIGIBILITY:
Inclusion Criteria:

* High-level athlete, enrolled in a Ministry-recognized Pôle
* Participant signed the informed consent form

Exclusion Criteria:

* Confirmed current overtraining syndrome
* Known pregnancy on inclusion
* Athlete using cardio-inhibitor or cardio-accelerator drugs

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: High-level athlete, enrolled in a Ministry-recognized Pôle
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Autonomic nervous system (ANS) activity | One year
  This ANS is mesured during the night using a spectral analysis of nocturnal heart rate variability.
Fatigue and physical training | One year
  Fatigue and physical training potetially due to overtraining, suspected based on a very significant, long-term worsening in performance

SECONDARY OUTCOMES:
kinetic of the ANS activity | Every 15 days (from the iclusion to one year)
  ANS is mesured during the night using a spectral analysis of nocturnal heart rate variability
orthostasis test | Every 15 days (from inclusion to one year)
  ANS activity measurements (RR variability) during active orthostasis transition on waking up in the morning
French Society of Sports Medicine questionnaire | Every 15 days (from inclusion to one year)
  The questionnaire was designed to detect early signs of overtraining. It includes 54 yes/no questions. Subjects who answer "yes" to more than 20 questions are considered at risk for overtraining.
POMS (Profile of Mood States) questionnaire | Every 3 months (from inclusion to inclusion)
Sleep quality questionnaire | Every 3 months (from inclusion to one year)
  The questionnaire is self-administered. It includes two parts. The first part consists of several questions regarding sleep during the previous night. The second part aims to evaluate the physical exertion load during the previous day's training session(s). Participants will fill one questionnaire/day for a whole week. Each questionnaire period must coincide with a training period (interseason, volume, intensity, or competition.)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ROCHE, MD PhD, Principal Investigator — CHU de Saint-Etienne; Xavier BIGARD, MD PhD, Study Chair — Institut de Recherche Biomédicales des Armées
Locations (8):
- France (8):
  - CH Albertville Moutiers, Albertville
  - CHU de Besançon, Besançon
  - Université Paris XIII, Bobigny
  - CHU de Grenoble, Grenoble
  - CHU de Pointe à Pitre, Pointe à Pitre
  - CNSN Centre médical de Prémanon, Prémanon
  - CHU de Saint-Etienne, Saint-Etienne
  - CREPS Toulouse Midi Pyrénées, Toulouse